CLINICAL TRIAL: NCT01692223
Title: Personal Genomics: A Safety Study Assessing the Effects of Receiving Genome Sequencing Results
Brief Title: A Safety Study Assessing the Effects of Receiving Genome Sequencing Results
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12-167
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: History of Cancer
Keywords: Personal genomics; Genome Sequencing Results; 12-167

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will be recruited from cohorts of patients whose DNA samples are being examined with WGS/WES as part of efforts to identify novel cancer susceptibility alleles. Participants will be derived from the following protocols: 09-068 and 96-051.

GROUPS / COHORTS (3):
- Unaffected Relatives: We will use a prospective, observational cohort design, we will invite a sample of individuals who have indicated willingness to be re-contacted for future studies (from existing protocols involving cancer survivors and their unaffected relatives employing mixed methods -qualitative interviews coupled with validated measures - to assess: the proportion of participants experiencing psychological distress from Whole genome/exome sequencing (WGS/WES) results.
  Interventions: Behavioral: qualitative interviews
- Pts with history of cancer: We will use a prospective, observational cohort design, we will invite a sample of individuals who have indicated willingness to be re-contacted for future studies (from existing protocols involving cancer survivors and their unaffected relatives employing mixed methods -qualitative interviews coupled with validated measures - to assess: the proportion of participants experiencing psychological distress from Whole genome/exome sequencing (WGS/WES) results.
  Interventions: Behavioral: qualitative interviews
- Participants whose genomes/exomes are not sequenced: We will also recruit an additional group of participants from the general public (with or without a cancer history) who have not had their genomes or exomes sequenced to participate in focus groups to inform us about their perceptions of the hypothetical utility of learning of incidental results from their genome or exomes. For our sampling purposes, this group of participants is referred to as the 'focus group participants (sample #3-hypothetical group)
  Interventions: Behavioral: qualitative interviews

INTERVENTIONS:
Behavioral: qualitative interviews — A week before the participants return to the clinic to learn of their results, the RSA will call each participant to complete the Hospital Anxiety & Depression Scale (HADS), revised Impact of Events Scale (IES-R), & a questionnaire about their health behaviors, to establish baseline distress levels & health behaviors. A week later, participants will return to the Clinical Genetics Service to review their results with the genetics provider & discuss resultant therapeutic & management recommendations for the participants & their relatives. A week later, the RSA will call each participant to complete the HADS, IES-R again, to establish the safety of receiving these results. Participants will also be asked to complete the revised Multidimensional Impact of Cancer Risk Assessment (MICRA) measure. The RSA will also invite participants to complete an in-depth telephone interview.
  Other Names: (Continued from Intervention Description) The RSA will call each participant to assess changes in health behavior and; service use at 3-,6- & 12-month timepoints after the results session. Distress; will also be re-assessed at 6 & 12-month timepoints after the results session.; The interviewer will call willing participants to complete an open-ended, in-depth; qualitative interview, approximately 3 months after their results session.

SUMMARY:
This study uses new methods called "genome sequencing" that allow the investigators to study part or all of a person's genome. The genome is the collection of all of a person's genes. Genes carry the instructions that our bodies need to develop and function. Genes are passed on from one generation to the next. Genome sequencing can study all of a person's genome (whole genome sequencing) or just parts of their genome (whole exome sequencing). In the study, the investigators refer to all these research methods as 'genome sequencing'. Genome sequencing typically shows a large number of gene changes, known as "variants." Some (but not all) of these genetic variants may be linked to increased risks of diseases other than cancer.

The purpose of this study is to learn what kinds of genetic variants the patient wants to learn about from their genome.

ELIGIBILITY:
Inclusion Criteria:

Cancer survivors (sample #1):

* Consented individuals with a personal history of cancer enrolled on protocols 09-068 or 96-051 who have indicated their interest in participating in future research or learning their results, defined as either:
* For samples #1-2: checking "yes" to the re-contact question in their consent form; or,
* checking "I wish to know these results" in their consent form.

Unaffected Relatives (sample #2):

* Consented individuals with no personal history of cancer enrolled on protocols 09-068 and 96-051 (parents or siblings of probands) who have indicated their interest in participating in future research or learning their results, defined as either:
* checking "yes" to the re-contact question in their consent form or,
* checking "I wish to know these results" in their consent form

Focus group participants (sample #3- hypothetical group):

* Individuals with or without a personal history of cancer

Exclusion Criteria:

* Non-English speakers; or,
* Individuals < 18 years of age; or
* Individuals unable to complete the follow-up assessments (e.g., unavailable to complete questionnaires over the 12-month study period).
* For samples #1-2: Individuals who indicate in their consent form that they do not want to
* checking "no" to the re-contact question in their consent form; or,
* checking "I prefer not to know these results" in their consent form
* Cases where it is unclear whether individuals' are interested in participating in future research or learning their results, defined as:
* Not answering the re-contact question in their consent form (i.e., left blank); or,
* Not answering the re-contact question because it did not exist in the version of the consent form that was originally signed (i.e., re-contact question missing).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from cohorts of patients whose DNA samples are being examined with WGS/WES as part of efforts to identify novel cancer susceptibility alleles. Participants will be derived from the following protocols: 09-068 and 96-051. We will also recruit an additional group of participants (up to 100) from the general public (with or without a cancer history) who have not had their genomes or exomes sequenced to participate in focus groups to inform us about their perceptions of the hypothetical utility of learning of incidental results from their genome or exomes.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-09; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Psychological distress | 2 years
  of receiving incidentally identified disease risk results from whole genome/exome sequencing. Safety is defined as no more than 20% of participants experiencing clinically meaningful levels of distress at 1 week follow-up, as measured by the Hospital Anxiety & Depression Scale (HADS; score > or = to 8 on the anxiety sub-scale). Patients will be considered evaluable for the primary outcome if they are not distressed at baseline and have completed the 1 week follow-up assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Robson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/